CLINICAL TRIAL: NCT03175549
Title: Medication Development for Protracted Abstinence in Alcoholism: Apremilast Versus Placebo
Brief Title: Medication Development in Alcoholism: Apremilast Versus Placebo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Scripps Research Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: U01AA025476 (NIH)
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Results first posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-08

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — apremilast; Sugars

STUDY DESIGN:
Intervention Model Description: Parallel Assignment, Double Blind, Randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apremilast (Otezla) (Active Comparator): Fixed oral dose of 90 mg/d following the standard titration for a total dosing duration of 14 days.
  Interventions: Drug: Apremilast
- Placebo (Placebo Comparator): Identical placebo pills taken orally for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apremilast — Fixed oral dose of 90 mg/d following the standard titration for a total dosing duration of 14 days.
  Other Names: Otezla
  Arms: Apremilast (Otezla)
Drug: Placebo — Identical placebo pills taken orally for 14 days
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The primary hypotheses under test are that alcohol dependent subjects treated with apremilast will report decreased craving for alcohol following alcohol exposure in the laboratory and report significantly less drinking under naturalistic conditions, than those treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers, 18-65 years of age
* Meets DSM-5 criteria for current alcohol use disorder of moderate or greater severity (AUD-MS)
* In the month prior to screening, reports drinking ≥ 21 standard drinks per week if male, ≥ 14 if female, with at least one heavy drinking day (≥ 5 males, ≥ 4 females) per week.
* Subjects will not be seeking treatment because the medication studies are not treatment trials, and to avoid exposing treatment-seekers to alcohol cues
* Subjects must be abstinent a minimum of 3 days (but not more than 7 days) prior to the human lab session
* Negative BAC and a CIWA score of < 9 at time of lab session to eliminate acute alcohol or withdrawal effects on dependent measures.
* In acceptable health in the judgment of the study physician, on the basis of interview, medical history, physical exam, EKG, routine urine and blood chemistry.
* Females with childbearing potential must have a negative pregnancy test on the screening, randomization, and lab session visits and agree to use effective birth control for the duration required by a given study.
* Able to provide informed consent and understand questionnaires and study procedure
* Willing to comply with the provisions of the protocol and take daily oral medication.

Exclusion Criteria:

* Active suicidal ideation, as systematically assessed with the Columbia Suicide Severity Rating Scale.
* Meets DSM-5 criteria for a major psychiatric disorder, including mood or anxiety disorders or substance use disorders other than alcohol or nicotine
* Has a urine drug screen (UDS) positive for substances of abuse other than alcohol.
* Significant medical disorders that will increase potential risk or interfere with study participation as determined by the study physician
* Known hypersensitivity to apremilast
* Treatment within the month prior to screening with (1) an investigational drug, (2) medications which may negatively interact with study medications, or (3) drugs that may influence study outcomes (e.g., disulfiram [Antabuse], naltrexone [ReVia], acamprosate [Campral], anticonvulsants, or antidepressants).
* Ongoing treatment with medications that may increase risk, including prescribed, over-the-counter, and herbal preparations, as determined by the study physician.
* Sexually active female subjects with childbearing potential who are pregnant, nursing, or refuse to use effective methods of birth control for the duration required by a specific protocol.
* No fixed domicile and/or no availability by home or mobile telephone
* History of hypersensitivity to the study drug or the ingredients.
* Failure to take double-blind medication as prescribed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Mason, Ph.D., Principal Investigator — The Scripps Research Institute
Locations (1):
- The Scripps Research Institute Pearson Center for Alcoholism and Addiction Research, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited for study participation at the Laboratory of Clinical Psychopharmacology at The Scripps Research Institute in La Jolla, CA from 11/01/2017-04/01/2020. Seventy-seven non-treatment seeking, paid volunteers signed informed consent, Fifty-one subjects were enrolled, and Forty-three subjects completed the study.
Pre-assignment Details: Twenty-six subjects were excluded from study participation, twenty-two did not meet admission criteria and four declined to participate.
Groups:
- Apremilast (Otezla): Fixed oral dose of 90 mg/d following standard titration for a total duration of 14 days.
- Placebo: Placebo pill taken orally for 14 days
  Placebo: Oral pill, 14 days
Period: Overall Study
Arm/Group | Apremilast (Otezla) | Placebo
Started | 26 | 25
Completed | 22 | 21
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 2 | 2
Not completed — Medication non-compliance | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo pill taken orally for 14 days
- Total: Total of all reporting groups
Arm/Group | Apremilast (Otezla) | Placebo | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.12 (13.9) | 43.3 (18.5) | 41.16 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 11 | 16 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 24 | 20 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 0 | 2
  White | 20 | 23 | 43
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 51
DSM-V symptom count [Mean (Standard Deviation); unit: Symptom count] | 6.58 (2.2) | 6.24 (2.4) | 6.41 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Craving to Drink
Description: Total Visual Analog Scale (VAS) scores of craving severity in response to in vivo alcohol cues. Higher scores indicate greater craving severity with a minimum score of 0 and a maximum score of 80.
Time Frame: 1 hour on the last day of dosing (Day 14)
Population: All subjects who completed cue exposure testing in the laboratory were included.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apremilast (Otezla) | Placebo
Number analyzed (Participants) | 21 | 20
score on a scale | 33.84 [14.03 to 53.73] | 28.31 [8.34 to 48.11]
Statistical Analysis 1: Comparison: Apremilast (Otezla) vs Placebo; Test type: Superiority; p = 0.36, Mixed Models Analysis — A priori threshold for significance was 0.05; Mean Difference (Final Values) = 5.53, 95% CI 2-sided [-10.22 to 29.38], Standard Error of Mean 10.10 — Standard error was calculated using bootstrap methods which is considered best for MEM

2. Secondary Outcome: Drinking
Description: Number of standard drinks per day using the Timeline Followback Interview (TLFB). Total number of alcoholic drinks consumed per day with a minimum value of 0 and an undetermined maximum value.
  Treatment effects on drinking were accessed during the 11 days of ad libidum and did not include the final three days of mandatory abstinence prior to cue reactivity testing on day 14 of dosing.
Time Frame: 11 days (Treatment effects on drinking were accessed during the 11 days of ad libidum and did not include the final three days of mandatory abstinence prior to cue reactivity testing on day 14 of dosing.)
Population: All subjects with post baseline drinking data were included.
Measure: Mean (Standard Error); unit: Drinks per day
Arm/Group | Apremilast (Otezla) | Placebo
Number analyzed (Participants) | 22 | 21
Drinks per day | 3.71 (0.82) | 3.92 (0.82)
Statistical Analysis 1: Comparison: Apremilast (Otezla) vs Placebo; Posted results show mean change in drinking for the drug group relative to placebo for each day of the 11 days of ad libidum drinking (Days 1-11) permitted during the 14 days (2 weeks) of medication; Test type: Superiority; p < 0.025, t-test, 2 sided; Slope = -0.067, Standard Error of Mean 0.030
Statistical Analysis 2: Comparison: Apremilast (Otezla) vs Placebo; Test type: Superiority; p = 0.025, Mixed Models Analysis; 473 daily observations within 43 individuals; Slope = -0.067, Standard Error of Mean 0.03 — The apremilast group showed a significantly more rapid reduction in drinks per day relative to placebo

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at all study visits, for an average duration of 4 weeks (2 weeks on drug, and 2 weeks post treatment).
Description: Adverse events, both serious and other, were documented at all study visits by the Medical Assistant on the adverse events case report form.
Arm/Group | Apremilast (Otezla) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 22/26 | 19/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apremilast (Otezla) (N=26) | Placebo (N=25)
Abdominal Pain (Gastrointestinal disorders) | 4 | 0
Diarrhea (Gastrointestinal disorders) | 9 | 4
Nausea (Gastrointestinal disorders) | 11 | 4
Hangover (General disorders) | 4 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Headache (Nervous system disorders) | 10 | 9
Somnolence (Nervous system disorders) | 7 | 3
Insomnia (Psychiatric disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-06-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT03175549/Prot_002.pdf
  • Statistical Analysis Plan (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT03175549/SAP_003.pdf
  • Informed Consent Form (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT03175549/ICF_004.pdf